CLINICAL TRIAL: NCT06507657
Title: Effect of Empagliflozin on Left Atrial Function in Adults at Risk for Heart Failure
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV-2023-32230
Record Dates: First submitted 2024-07-11; First posted 2024-07-18 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Hypertension; Cardiovascular Diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: placebo-controlled, double-blinded, randomized pilot study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Drug: empagliflozin
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo tablet

INTERVENTIONS:
Drug: empagliflozin — intake of a 10mg empagliflozin oral tablet
  At visit 1, after randomization, participants will be provided with bottles containing enough study pills for 3 months duration at 1 tablet daily. Participants will start the study drug on the morning following Visit 1. At the 3 month follow up visit, participants will be provided with enough study pills to complete the remaining 6 months of the study.
  Arms: Experimental group
Drug: Placebo tablet — intake a placebo oral tablet
  At visit 1, after randomization, participants will be provided with bottles containing enough study pills for 3 months duration at 1 tablet daily. Participants will start the study drug on the morning following Visit 1. At the 3 month follow up visit, participants will be provided with enough study pills to complete the remaining 6 months of the study.
  Arms: Placebo group

SUMMARY:
Sodium-glucose cotransporter 2 inhibitors (SGLT2i) reduce CVD events, including incident HF. SGLT2 is a glucose transport protein in the kidneys. Inhibition of this protein results in glucosuria and lower serum blood sugar. The SGLT2i medications were initially approved to treat type 2 diabetes (T2D). In 2015, Zinman et al. published the first large randomized clinical trial (RCT) demonstrating a lower composite CVD outcome in adults with T2D treated with empagliflozin compared to placebo (HR 0.85, 95% CI 0.74-0.99). In the specific case of empagliflozin, the hazard ratio was 0.75 (95% CI 0.65-0.86) for HFrEF 8 and 0.79 (95% CI 0.69-0.90) for HFpEF using a treatment dose of 10mg daily.

The purpose of this placebo-controlled, double-blinded, randomized pilot study is to investigate the effect of empagliflozin on left atrial (LA) function in 80 patients who are at risk for heart failure. Participants will be randomized 1:1 to either intake of a 10mg empagliflozin oral tablet or a matching placebo once daily.

ELIGIBILITY:
Inclusion Criteria:

* Age >60 years of age
* Clinical diagnosis of hypertension
* Body mass index ≥30kg/m2
* We will screen for participants with an echocardiogram within 60 days of the baseline visit

Exclusion Criteria:

* Female participants who are pregnant, lactating, or of child bearing potential
* History of type 1 or type 2 diabetes mellitus by medical history or hemoglobin A1c >7.0% at Visit 1
* Clinical diagnosis of HFpEF or HFrEF by participant self-report or documented in the electronic health record
* Any LVEF measure of ≤40% on past echocardiogram
* Moderate or severe valve disease on echocardiogram
* History of genitourinary infection
* eGFR <60 ml/min/1.73 m2 at Visit 1
* Current treatment with SGLT2 inhibitor, GLP1 agonist, or DPP4 inhibitors
* Participants in whom coronary revascularization by either PCI or bypass surgery is being contemplated within 6 months, or who have undergone revascularization in the prior 2 months
* Significant allergy or known intolerance to SGLT2 inhibitors or any ingredient in the formulations
* Participants currently experiencing any clinically significant or unstable medical condition that might limit their ability to complete the study, or to comply with the requirements of the protocol, including: dermatologic disease, hematological disease, pulmonary disease, hepatic disease, gastrointestinal disease, genitourinary disease, endocrine disease, neurological disease, and psychiatric disease
* Any malignancy not considered cured (except basal cell carcinoma of the skin). A participant is considered cured if there has been no evidence of cancer recurrence for the 5 years prior to screening
* Participants who have participated in studies of an investigational drug or device within 30 days prior to the screening visit
* Inadequate quality echocardiographic images
* Unstable coronary syndromes
* Major surgery (major according to the investigator's assessment) performed within 90 days prior to Visit 1 or scheduled major elective surgery within 90 days after Visit 1.
* Non-English speaking individuals

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2029-01-15 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
change in LA function | 9 months
  LA function will be quantified by assessing LA reservoir, conduit, and contractile strain with 2DE at baseline and 9 months.

SECONDARY OUTCOMES:
change in left ventricular ejection fraction | 9 months
change in global longitudinal strain | 9 months
change in mass (indexed to body surface area) | 9 months
change in E/e' ratio | 9 months
change in plasma protein levels: DLK-1 (protein delta homolog 1) | 9 months
change in plasma protein levels: GDF15 (growth differentiating factor 15) | 9 months
change in plasma protein levels: Spondin-1 | 9 months
change in plasma protein levels: IGBPF-7 | 9 months
change in plasma protein levels: THBS-2 (thrombospondin 2) | 9 months
change in plasma protein levels: IGFBP-1 (insulin-like binding factor protein 1) | 9 months
change in plasma protein levels: FABP-4 (fatty acid-binding protein 4) | 9 months
change in plasma protein levels: CCL16 (C-C motif chemokine 16) | 9 months
change in cardiovascular disease biomarker C-reactive protein (CRP) | 3 months and 9 months
change in cardiovascular disease biomarker Troponin | 3 months and 9 months
change in cardiovascular disease biomarker NT-proBNP | 3 months and 9 months
changes in blood pressure ration | 1, 3 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Van't Hof, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States